CLINICAL TRIAL: NCT03954340
Title: BestBrain Evaluation of Cognitive Memory & Executive-Function (BECOME)
Brief Title: BestBrain Evaluation of Cognitive Memory & Executive-Function
Acronym: BECOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BestBrain Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIP001
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Mild Cognitive Impairment
Keywords: MCI; Early AD
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Subjects will undergo either EEG NFB treatment with the iRemember System or a sham treatment
Who Masked: Participant, Care Provider, Investigator
Masking Description: all will be blinded to sham or treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 iRemember Treatment (Active Comparator): Subjects randomized to this arm of the study will undergo 20 EEG NFB treatments with the iRemember System for the treatment of MCI
  Interventions: Device: iRemember Neurofeedback (NFB)
- 2 Sham Treatment (Sham Comparator): Subjects randomized to this arm of the study will undergo 20 SHAM treatments
  Interventions: Device: iRemember Neurofeedback (NFB)

INTERVENTIONS:
Device: iRemember Neurofeedback (NFB) — Neurofeedback (NFB) is a treatment technique based on learning with operant conditioning, in which a feedback (or a reward) is given in proportion with the desired physiological activity in order to improve cognition and/or behavior. This research will focus on EEG-NF where electrical activity measured with EEG serves as the physiological activity to be influenced.
  EEG-NFB has been successfully used as a clinical tool for over 40 years treating various disorders from Autism , ADHD , Epilepsy , OCD and depression Electroencephalography (EEG) equipment is used to measure the electrical activity representing the neuronal activity of different parts of the brain.
  During the treatment, electrode(s) are placed in predetermined location. Audio and visual rewards are given when the activity is measured to be within the desired frequency range.
  Other Names: EEG NFB

SUMMARY:
This study is intended 1. To quantify the effects of the iRemember personalized EEG-NFB therapy on working memory and executive functions in subjects with MCI by calculating the percentage of change in the Neurotrax tests performed prior to and after the treatment, and compare the results between the active treatment and placebo cohorts

DETAILED DESCRIPTION:
By using the BestBrain iRemember EEG-NFB System, subjects within the "treatment" arm of this clinical investigation will show improvement in working memory, executive functions and general improvement in daily life based on standard accepted cognitive tests such as the Neurotrax and Kielhfner questionnaire. This hypothesis will be accepted or rejected based on the statistical analysis of the data collected .

Subjects will be randomized either to the treatment or placebo groups. Each subject will undergo an initial and final assessment using NeuroTrax and specified questionnaires prior to and after 20 treatments. The first sessions will be dedicated to subject evaluation. Each subject will undergo either a neurofeedback (NFB) or sham treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 50-80 years
2. Subjects diagnosed with MCI, according to the ICD-10 criteria.
3. MoCA score 18 to 25
4. Ability to operate a computer mouse and keyboard as evaluated by the clinician.
5. Agreement to participate in approximately 12 weeks during the study.
6. Normal to near-normal vision and hearing with correction as needed (e.g. corrective lenses, hearing aid).
7. Fluent in Hebrew
8. Willing to participate twice a week for treatments

Exclusion Criteria:

1. Participation in a clinical trial with any investigational agent within 6 months prior to study enrollment
2. Subjects with one or more of the following disorders in their medical files: psychotic disorder, currently active depression, with a history of bipolar disorder, adjustment disorder, somataform disorder, anxiety disorder OCD, PTSD. (following the Axis-1 disorders listed in the ICD-10)
3. Alcoholism or drug addiction as defined by ICD-10 within last 5 years (addicted more than one year and or in remission less than 3 years) or severe sleep deprivation
4. Subjects with personal history of a clinically defined neurological/psychiatric disorder including (but not limited to): epilepsy, dementia, clinical stroke (hemiparesis, hemianopsia) , substance abuse, extra pyramidal disorders like parkinson etc) , major head trauma, multiple sclerosis; or personal history of previous neurosurgery or head trauma that resulted in loss of consciousness; use of any medication with the aim to improve cognition (cholinesterase inhibitors).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Improvement to Memory | 3-4 months
  Improvement in memory based on evaluation before and after treatment with the iRemember EEG NFB System (greater than in subjects who received SHAM treatments)
Improvement to Executive Functions | 3-4 months
  Improvement to Executive Functions based on evaluation before and after treatment with the iRemember EEG NFB System (greater than in subjects who received SHAM treatments)
Improvement to Every Day Functionality | 3-4 months
  Improvement Every Day Functionality based on evaluation before and after treatment with the iRemember EEG NFB System (greater than in subjects who received SHAM treatments)

CONTACTS AND LOCATIONS:
Locations (1):
- Clalit Health Services, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No